CLINICAL TRIAL: NCT02476006
Title: A Multi-country, Multicenter, Single-arm, Open-label Study to Document the Safety, Tolerability and Effect of Alirocumab on Atherogenic Lipoproteins in High Cardio-vascular Risk Patients With Severe Hypercholesterolemia Not Adequately Controlled With Conventional Lipid-modifying Therapies
Brief Title: Safety, Tolerability, and Effect of Alirocumab in High Cardiovascular Risk Patients With Severe Hypercholesterolemia Not Adequately Controlled With Conventional Lipid-modifying Therapies (ODYSSEY APPRISE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS14245; 2015-000620-28 (EudraCT Number); U1111-1163-0984 (Other: UTN)
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Ezetimibe; Atorvastatin; Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- Alirocumab (Experimental): Participants received Alirocumab 150 milligram (mg) subcutaneously (SC) once every two weeks (Q2W) or 75 mg SC Q2W added to stable LMT up to a maximum of 120 weeks. Alirocumab dose was either up-titrated from 75 to 150 mg Q2W or down-titrated from 150 to 75 mg Q2W, based on Investigator judgment and treatment response.
  Interventions: Drug: ALIROCUMAB SAR236553 (REGN727); Drug: placebo (for injection training only); Drug: ezetimibe; Drug: atorvastatin; Drug: rosuvastatin; Drug: simvastatin

INTERVENTIONS:
Drug: ALIROCUMAB SAR236553 (REGN727) — Pharmaceutical form:solution Route of administration: subcutaneous
  Other Names: Praluent®
Drug: placebo (for injection training only) — Pharmaceutical form:solution Route of administration: subcutaneous
Drug: ezetimibe — Pharmaceutical form:capsule Route of administration: oral
Drug: atorvastatin — Pharmaceutical form:tablet Route of administration: oral
Drug: rosuvastatin — Pharmaceutical form:tablet Route of administration: oral
Drug: simvastatin — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

To provide participants with severe hypercholesterolemia at risk for subsequent cardiovascular (CV) events and not adequately controlled with currently available lipid-modifying therapy (LMT) access to alirocumab ahead of commercial availability and to document the overall safety and tolerability of alirocumab in this participant population.

Secondary Objectives:

To document the effect of alirocumab on low-density lipoprotein cholesterol (LDL-C) levels as well as non-high-density lipoprotein cholesterol (non-HDL-C), total cholesterol (total-C), high-density lipoprotein cholesterol (HDL-C), and triglyceride (TG) levels after 12 weeks of treatment.

To document participant's acceptability of self-injection (Self Injection Assessment Questionnaire, SIAQ).

DETAILED DESCRIPTION:
The study duration included a screening period of up to 3 weeks, a treatment period of a minimum of 12 weeks and up to a maximum of 120 weeks (30 months), and at least 2 weeks after the last study treatment injection.

ELIGIBILITY:
Inclusion criteria:

Either A, B, C, D, or E below and not adequately controlled with a maximally tolerated dose of statin with or without other LMTs, all at stable doses for at least 4 weeks prior to the screening visit (Week-3):

A. Participants suffering from heterozygous familial hypercholesterolemia (heFH) with LDL-C concentrations greater than or equal to (>=)160 mg/dL (4.14 millimoles per liter [mmol/L]) despite treatment.

B. Participants suffering from heFH with LDL-C concentrations >=130 mg/dL (3.36 mmol/L) despite treatment and two or more CV risk factors among this list:

* LDL-C greater than (>) 250 milligrams per deciliter (mg/dL) (6.46 mmol/L) at the time of the familial hypercholesterolemia (FH) diagnosis (before treatment).
* Family history of premature-onset coronary heart disease (CHD; first-degree male relative with onset before age 55 years; first-degree female relative with onset before age 65 years).
* Metabolic syndrome.
* HDL-C less than (<) 40 mg/dL (1.03 mmol/L).
* Hypertension (blood pressure >140/90 mmHg or drug treatment).
* Lipoprotein a (Lp[a]) >=50 mg/dL (1.78 µmol/L).
* Tendon xanthoma.

C. Participants suffering from heFH with LDL-C concentrations >=130 mg/dL (3.36 mmol/L) despite treatment and one of the following characteristics:

* Established CHD or other cardiovascular disease (CVD; history of acute myocardial infarction, ischemic stroke, peripheral arterial disease, coronary or peripheral arterial revascularization, stable or unstable angina, transient ischemic attack, carotid artery stenosis >=50 percent (%), or aortic abdominal aneurysm).
* Drug-treated type 2 diabetes mellitus or type 1 with target organ damage.
* Family history of first- or second-degree relative with very premature onset CHD (first- or second-degree male relative with onset before age 45; first- or second-degree female relative with onset before age 55).

D. Non-FH participants suffering from established CHD or other CVD (history of acute myocardial infarction (MI), ischemic stroke, peripheral arterial disease, coronary or peripheral arterial revascularization, stable or unstable angina, transient ischemic attack, carotid artery stenosis >=50%, or aortic abdominal aneurysm) and with LDL-C concentrations >=130 mg/dL (3.36 mmol/L).

E. Participants suffering from progressive CVD (coronary artery disease, or peripheral arterial occlusive disease or cerebrovascular disease as documented clinically or by imaging techniques, with a subsequent CV event [acute MI, ischemic stroke, ischemia-driven revascularization, unstable angina, transient ischemic attack] occurring despite stable doses of maximally tolerated LMT) with LDL-C concentrations >=100 mg/dL (2.59 mmol/L).

Exclusion criteria:

Not on a stable dose of LMT (including statin) for at least 4 weeks prior to the screening visit (Week -3) and from screening to enrollment.

Use of a fibrate other than fenofibrate within 4 weeks of the screening visit (Week-3) or between screening and enrollment.

Daily doses above atorvastatin 80 mg, rosuvastatin 40 mg, or simvastatin 40 mg (except for participants on simvastatin 80 mg for more than one year, who were eligible).

Use of statin other than simvastatin, atorvastatin, or rosuvastatin prior to the screening visit (Week-3) or between screening and enrollment, except when there was a documented reason for intolerance to the above mentioned potent statins (in which case the use of a different statin was allowed).

Fasting serum TG >400 mg/dL (>4.52 mmol/L) at the screening visit (Week -3). Uncontrolled hypertension (>180 mmHg systolic and/or >110 mmHg diastolic at randomization visit).

New York Heart Association Class III or IV congestive heart failure persisting despite treatment.

History of hemorrhagic stroke. Liver transaminases >3 times the upper limit of normal. Laboratory evidence of current hepatitis B or C infection. Creatine kinase >3 times the upper limit of normal. Estimated glomerular filtration rate <30 mL/min/1.73 m^2. Pregnant or breastfeeding woman or with childbearing potential without appropriate contraception.

Male participant with a female partner of childbearing potential not protected by a highly-effective method(s) of birth control.

Participants eligible for enrollment into an ongoing clinical study of alirocumab conducted at the same investigational site.

Hypersensitivity to alirocumab or any of the excipients.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 998 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (153):
- Austria (9):
  - Investigational Site Number 040001, Graz
  - Investigational Site Number 040008, Innsbruck
  - Investigational Site Number 040005, Linz
  - Investigational Site Number 040006, Linz
  - Investigational Site Number 040003, Vienna
  - Investigational Site Number 040002, Vienna
  - Investigational Site Number 040004, Vienna
  - Investigational Site Number 040007, Vienna
  - Investigational Site Number 040010, Vienna
- Belgium (18):
  - Investigational Site Number 056005, Aalst
  - Investigational Site Number 056018, Antwerp
  - Investigational Site Number 056008, Arlon
  - Investigational Site Number 056013, Bruges
  - Investigational Site Number 056010, Brussels
  - Investigational Site Number 056003, Brussels
  - Investigational Site Number 056006, Charleroi
  - Investigational Site Number 056007, Edegem
  - Investigational Site Number 056019, Genk
  - Investigational Site Number 056001, Ghent
  - Investigational Site Number 056017, Ghent
  - Investigational Site Number 056002, Haine-Saint-Paul
  - Investigational Site Number 056015, Kortrijk
  - Investigational Site Number 056009, La Louvière
  - Investigational Site Number 056004, Leuven
  - Investigational Site Number 056014, Liège
  - Investigational Site Number 056011, Overpelt
  - Investigational Site Number 056016, Roeselare
- Canada (26):
  - Investigational Site Number 124018, Calgary
  - Investigational Site Number 124015, Cambridge
  - Investigational Site Number 124002, Chicoutimi
  - Investigational Site Number 124027, Coquitlam
  - Investigational Site Number 124025, Edmonton
  - Investigational Site Number 124017, Halifax
  - Investigational Site Number 124013, Hamilton
  - Investigational Site Number 124008, London
  - Investigational Site Number 124026, Maple Ridge
  - Investigational Site Number 124020, Montreal
  - Investigational Site Number 124022, Montreal
  - Investigational Site Number 124032, Mount Pearl
  - Investigational Site Number 124005, Ottawa
  - Investigational Site Number 124024, Peterborough
  - Investigational Site Number 124003, Québec
  - Investigational Site Number 124019, Saint-Charles-Borromée
  - Investigational Site Number 124007, Sarnia
  - Investigational Site Number 124001, Sherbrooke
  - Investigational Site Number 124030, Smiths Falls
  - Investigational Site Number 124023, Toronto
  - Investigational Site Number 124014, Toronto
  - Investigational Site Number 124028, Trois-Rivières
  - Investigational Site Number 124011, Vancouver
  - Investigational Site Number 124012, Victoria
  - Investigational Site Number 124031, Winnipeg
  - Investigational Site Number 124009, Woodstock
- Czechia (4):
  - Investigational Site Number 203004, Brno
  - Investigational Site Number 203002, Hradec Králové
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203005, Uherské Hradiště
- Denmark (3):
  - Investigational Site Number 208003, Aalborg
  - Investigational Site Number 208001, Esbjerg
  - Investigational Site Number 208002, Roskilde
- Finland (2):
  - Investigational Site Number 246003, Turku
  - Investigational Site Number 246001, Varkaus
- France (47):
  - Investigational Site Number 250027, Amiens
  - Investigational Site Number 250034, Auxerre
  - Investigational Site Number 250016, Avignon
  - Investigational Site Number 250021, Bayonne
  - Investigational Site Number 250030, Bobigny
  - Investigational Site Number 250045, Bordeaux
  - Investigational Site Number 250049, Brest
  - Investigational Site Number 250054, Bron
  - Investigational Site Number 250015, Caen
  - Investigational Site Number 250047, Clermont-Ferrand
  - Investigational Site Number 250013, Corbeil-Essonnes
  - Investigational Site Number 250032, Coudray
  - Investigational Site Number 250002, Dijon
  - Investigational Site Number 250040, Dijon
  - Investigational Site Number 250012, Grenoble
  - Investigational Site Number 250038, Grenoble
  - Investigational Site Number 250033, Jossigny
  - Investigational Site Number 250035, Le Chesnay
  - Investigational Site Number 250036, Lens
  - Investigational Site Number 250042, Lille
  - Investigational Site Number 250004, Lille
  - Investigational Site Number 250037, Limoges
  - Investigational Site Number 250057, Lyon
  - Investigational Site Number 250028, Marseille
  - Investigational Site Number 250048, Marseille
  - Investigational Site Number 250024, Montpellier
  - Investigational Site Number 250006, Nantes
  - Investigational Site Number 250022, Nantes
  - Investigational Site Number 250017, Nice
  - Investigational Site Number 250039, Nîmes
  - Investigational Site Number 250014, Paris
  - Investigational Site Number 250041, Paris
  - Investigational Site Number 250026, Paris
  - Investigational Site Number 250044, Paris
  - Investigational Site Number 250001, Paris
  - Investigational Site Number 250051, Pessac
  - Investigational Site Number 250011, Poitiers
  - Investigational Site Number 250031, Poitiers
  - Investigational Site Number 250010, Reims
  - Investigational Site Number 250008, Rennes
  - Investigational Site Number 250018, Rouen
  - Investigational Site Number 250023, Saint-Mandé
  - Investigational Site Number 250025, Toulouse
  - Investigational Site Number 250046, Toulouse
  - Investigational Site Number 250007, Tours
  - Investigational Site Number 250019, Vénissieux
  - Investigational Site Number 250050, Vichy
- Germany (2):
  - Investigational Site Number 276001, Berlin
  - Investigational Site Number 276003, Magdeburg
- Greece (3):
  - Investigational Site Number 300003, Ampelokipoi
  - Investigational Site Number 300002, Ioannina
  - Investigational Site Number 300001, Kallithea
- Hungary (4):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348002, Debrecen
  - Investigational Site Number 348004, Pécs
  - Investigational Site Number 348003, Szeged
- Poland (5):
  - Investigational Site Number 616005, Gdansk
  - Investigational Site Number 616003, Krakow
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616004, Olsztyn
  - Investigational Site Number 616002, Warsaw
- Romania (3):
  - Investigational Site Number 642-003, Bucharest
  - Investigational Site Number 642-002, Iași
  - Investigational Site Number 642-001, Timișoara
- Slovakia (3):
  - Investigational Site Number 703003, Bratislava
  - Investigational Site Number 703002, Bratislava
  - Investigational Site Number 703001, Košice
- Investigational Site Number 705001, Maribor, Slovenia
- Spain (18):
  - Investigational Site Number 724009, Alicante
  - Investigational Site Number 724011, Alicante
  - Investigational Site Number 724003, Córdoba
  - Investigational Site Number 724012, Donostia / San Sebastian
  - Investigational Site Number 724014, Donostia / San Sebastian
  - Investigational Site Number 724019, Elche
  - Investigational Site Number 724017, Galdakao
  - Investigational Site Number 724020, Inca
  - Investigational Site Number 724001, L'Hospitalet de Llobregat
  - Investigational Site Number 724007, Las Palmas de Gran Canaria
  - Investigational Site Number 724004, Madrid
  - Investigational Site Number 724008, Madrid
  - Investigational Site Number 724010, Madrid
  - Investigational Site Number 724005, Málaga
  - Investigational Site Number 724002, Santiago de Compostela
  - Investigational Site Number 724006, Valencia
  - Investigational Site Number 724016, Valencia
  - Investigational Site Number 724015, Valladolid
- Switzerland (5):
  - Investigational Site Number 756005, Baden
  - Investigational Site Number 756002, Olten
  - Investigational Site Number 756004, Reinach
  - Investigational Site Number 756003, Sankt Gallen
  - Investigational Site Number 756001, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Cefalu AB, Garbelotto R, Mombelli G, Pirro M, Rubba P, Arca M, Borghi C, Bonomo K, Gonnelli S, Massaroni K, Tirone G, Averna M; ODYSSEY APPRISE Study Italian Investigators. A subgroup analysis of the ODYSSEY APPRISE study: Safety and efficacy of alirocumab in the Italian cohort. Nutr Metab Cardiovasc Dis. 2022 Nov;32(11):2638-2646. doi: 10.1016/j.numecd.2022.07.020. Epub 2022 Aug 9. PMID 36064689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 156 sites in 17 countries. A total of 1305 participants were screened between 23-June-2015 to 27-December 2016, of whom 307 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: A total of 998 participants were enrolled in the study.
Groups:
- Alirocumab: Participants received Alirocumab 150 milligram (mg) subcutaneously (SC) once every two weeks (Q2W) or 75 mg SC Q2W added to stable lipid modifying therapies (LMT) up to a maximum of 120 weeks. Alirocumab dose was either up-titrated from 75 to 150 mg Q2W or down-titrated from 150 to 75 mg Q2W, based on Investigator judgment and treatment response.
Period: Overall Study
Arm/Group | Alirocumab
Started | 998
Treated | 994
Completed | 878
Not Completed | 120
Not completed — Death | 4
Not completed — Lack of treatment efficacy | 2
Not completed — Pregnancy | 1
Not completed — Participant did not wish to continue | 39
Not completed — Adverse Event | 41
Not completed — Poor compliance to study protocol | 3
Not completed — Sponsor decision | 6
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 5
Not completed — Study ended treatment not available | 4
Not completed — Switched to commercial drug | 4
Not completed — Excluded from study | 1
Not completed — Protocol Violation | 1
Not completed — Enrolled but not treated | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population that included all participants who had signed the informed consent form (ICF) and who had received at least one dose or partial dose of alirocumab.
Groups:
- Alirocumab: Participants received Alirocumab 150 mg SC Q2W or 75 mg SC Q2W added to stable LMT up to a maximum of 120 weeks. Alirocumab dose was either up-titrated from 75 to 150 mg Q2W or down-titrated from 150 to 75 mg Q2W, based on Investigator judgment and treatment response.
Arm/Group | Alirocumab
Number analyzed (Participants) | 994
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 369
  Male | 625
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 969
  Black | 10
  Asian/Oriental | 6
  Multiracial | 1
  Other | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Treatment-emergent AEs (TEAEs) were defined as AEs that that developed or worsened or became serious during the TEAE period (time from the first injection of study drug up to the day of the last injection of study drug + 14 days). A Serious Adverse Event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From first injection of investigational medicinal product (IMP) up to 2 weeks after last dose of study drug (Week 120)
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab
Number analyzed (Participants) | 994
percentage of participants
  Any TEAE | 71.6
  Any treatment emergent SAE | 16.2
  Any TEAE leading to death | 0.2
  Any TEAE leading to treatment discontinuation | 4.5

2. Secondary Outcome: Percent Change From Baseline in Calculated Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: Calculated LDL-C values were obtained using the Friedewald formula. Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/5]). Baseline value was defined as the last observation before the first dose of the treatment.
Time Frame: Baseline, Week 12
Population: Analysis was performed on modified intent-to-treat population (mITT): all enrolled participants who received at least one dose or part of a dose of alirocumab and had an evaluable efficacy endpoint during the efficacy treatment period (defined as time period from the first injection of alirocumab up to the day of last injection +21 days).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percent change | -54.84 (20.06)

3. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 12
Description: LDL-Cholesterol was calculated using the Friedewald formula. Percentage of participants who reached calculated LDL-C <100 mg/dL (2.59 mmol/L) at week 12 were reported.
Time Frame: At Week 12
Population: Analysis was performed on mITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percentage of participants | 74.6 [71.7 to 77.4]

4. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 12
Description: LDL-Cholesterol was calculated using the Friedewald formula. Percentage of participants who reached calculated LDL-C <70 mg/dL (1.81 mmol/L) at week 12 were reported.
Time Frame: At Week 12
Population: Analysis was performed on mITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percentage of participants | 50.2 [46.9 to 53.4]

5. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) and/or >=50% Reduction From Baseline in LDL-C at Week 12
Description: LDL-Cholesterol was calculated using the Friedewald formula. Percentage of participants who reached LDL-C <70 mg/dL at Week 12 and/or >=50% reduction from baseline in LDL-C at Week 12 are reported.
Time Frame: At Week 12
Population: Analysis was performed on mITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percentage of participants | 69.1 [66.0 to 72.0]

6. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Description: Baseline value was defined as the last observation before the first dose of the treatment.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percent change | -45.89 (35.82)

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 12
Description: Baseline value was defined as the last observation before the first dose of the treatment.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percent change | -38.28 (15.20)

8. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol at Week 12
Description: Baseline value was defined as the last observation before the first dose of the treatment.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percent change | 4.37 (17.29)

9. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Description: Baseline value was defined as the last observation before the first dose of the treatment.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alirocumab
Number analyzed (Participants) | 921
percent change | -8.28 (33.99)

10. Secondary Outcome: Assessment of Participant's Acceptability of Self-Injection Using Self Injection Assessment Questionnaire (SIAQ): Feeling About Injections, Self Confidence, Satisfaction With Self-Injections
Description: Pre-SIAQ: self-completed before first self-injection & Post-SIAQ: self-completed after self-injection. Pre-SIAQ consisted of 7 items grouped into 3 domains:feelings about injections,self-confidence & satisfaction with self-injection. Post-SIAQ consisted of 21 items grouped into 6 domains:feelings about injections,self-image,self-confidence,injection-site reactions,ease of use & satisfaction with self-injection. Participants rated each item on 5-point (or 6-point) semantic Likert-type scale, where lower numbers indicate a worse experience. Item scores were transformed to obtain a score ranging from 0 (worst experience) to 10 (best experience). Transformed scores for items contributing to a domain were then averaged into a domain score. Each domain score ranges from 0 (worst experience) to 10 (best experience), higher score=better acceptability. Domain scores common to the Pre & Post SIAQ were analyzed on participants belonging to Pre & Post-SIAQ population and are reported.
Time Frame: Baseline (Pre-SIAQ), Week 4, Week 8, Week 12, Week 24, Week 48, Week 72, Week 96
Population: Pre and Post-SIAQ population: participants from the safety population who self-injected the training injection & completed a Pre-SIAQ before first self-injection, who self-injected study drug at least once during the study and completed a Post-SIAQ. Here, number analyzed = participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alirocumab
Number analyzed (Participants) | 952
units on a scale
  Feelings about injections: Baseline | 8.6 (1.8)
  Feeling about injections: Week 4: number analyzed (Participants) | 909
  Feeling about injections: Week 4 | 9.1 (1.4)
  Feeling about injections: Week 8: number analyzed (Participants) | 894
  Feeling about injections: Week 8 | 9.1 (1.4)
  Feeling about injections: Week 12: number analyzed (Participants) | 847
  Feeling about injections: Week 12 | 9.2 (1.4)
  Feeling about injections: Week 24: number analyzed (Participants) | 668
  Feeling about injections: Week 24 | 9.2 (1.4)
  Feeling about injections: Week 48: number analyzed (Participants) | 547
  Feeling about injections: Week 48 | 9.2 (1.4)
  Feeling about injections: Week 72: number analyzed (Participants) | 423
  Feeling about injections: Week 72 | 9.2 (1.4)
  Feeling about injections: Week 96: number analyzed (Participants) | 343
  Feeling about injections: Week 96 | 9.3 (1.3)
  Self confidence: Baseline: number analyzed (Participants) | 943
  Self confidence: Baseline | 6.9 (2.4)
  Self Confidence: Week 4: number analyzed (Participants) | 905
  Self Confidence: Week 4 | 8.0 (2.1)
  Self Confidence: Week 8: number analyzed (Participants) | 889
  Self Confidence: Week 8 | 8.1 (2.0)
  Self Confidence: Week 12: number analyzed (Participants) | 844
  Self Confidence: Week 12 | 8.1 (1.9)
  Self Confidence: Week 24: number analyzed (Participants) | 666
  Self Confidence: Week 24 | 8.0 (2.1)
  Self Confidence: Week 48: number analyzed (Participants) | 548
  Self Confidence: Week 48 | 8.1 (2.1)
  Self Confidence: Week 72: number analyzed (Participants) | 420
  Self Confidence: Week 72 | 8.3 (2.0)
  Self Confidence: Week 96: number analyzed (Participants) | 340
  Self Confidence: Week 96 | 8.4 (2.0)
  Satisfaction with self injection: Baseline: number analyzed (Participants) | 918
  Satisfaction with self injection: Baseline | 7.2 (2.5)
  Satisfaction with self-injections: Week 4: number analyzed (Participants) | 906
  Satisfaction with self-injections: Week 4 | 8.5 (1.6)
  Satisfaction with self-injections: Week 8: number analyzed (Participants) | 889
  Satisfaction with self-injections: Week 8 | 8.7 (1.6)
  Satisfaction with self-injections: Week 12: number analyzed (Participants) | 842
  Satisfaction with self-injections: Week 12 | 8.7 (1.6)
  Satisfaction with self-injections: Week 24: number analyzed (Participants) | 667
  Satisfaction with self-injections: Week 24 | 8.6 (1.8)
  Satisfaction with self-injections: Week 48: number analyzed (Participants) | 542
  Satisfaction with self-injections: Week 48 | 8.7 (1.5)
  Satisfaction with self-injections: Week 72: number analyzed (Participants) | 418
  Satisfaction with self-injections: Week 72 | 8.8 (1.7)
  Satisfaction with self-injections: Week 96: number analyzed (Participants) | 338
  Satisfaction with self-injections: Week 96 | 8.8 (1.4)

11. Secondary Outcome: Assessment of Participant's Acceptability of Self-Injection Using Self Injection Assessment Questionnaire (SIAQ): Self Image, Injection-Site Reactions, Ease of Use
Description: SIAQ: contained 2 modules: Pre-SIAQ and Post-SIAQ. Post-SIAQ: self-completed after self-injection. Post-SIAQ consisted of 21 items grouped into 6 domains: feelings about injections, self-image, self-confidence, injection-site reactions, ease of use & satisfaction with self-injection. Participants rated each item on 5-point (or 6-point) semantic Likert-type scale, where lower numbers indicated a worse experience. Item scores were transformed to obtain a score ranging from 0 (worst experience) to 10 (best experience) for each item. Transformed scores for items contributing to a domain were then averaged into a domain score. Each domain score ranges from 0 (worst experience) to 10 (best experience), higher score=better acceptability. Domain scores which are not in common with Pre-SIAQ were analyzed on the Post-SIAQ population and are reported here.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 48, Week 72, Week 96
Population: POST-SIAQ population: participants from safety population who self-injected at least once during the study and completed a POST-SIAQ regardless of completion of PRE-SIAQ. Here, number analyzed = participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alirocumab
Number analyzed (Participants) | 979
units on a scale
  Self Image: Week 4: number analyzed (Participants) | 929
  Self Image: Week 4 | 9.4 (1.4)
  Self Image: Week 8: number analyzed (Participants) | 915
  Self Image: Week 8 | 9.4 (1.4)
  Self Image: Week 12: number analyzed (Participants) | 866
  Self Image: Week 12 | 9.4 (1.4)
  Self Image: Week 24: number analyzed (Participants) | 682
  Self Image: Week 24 | 9.3 (1.5)
  Self Image: Week 48: number analyzed (Participants) | 560
  Self Image: Week 48 | 9.4 (1.4)
  Self Image: Week 72: number analyzed (Participants) | 433
  Self Image: Week 72 | 9.3 (1.5)
  Self Image: Week 96: number analyzed (Participants) | 349
  Self Image: Week 96 | 9.4 (1.4)
  Injection-site reactions: Week 4: number analyzed (Participants) | 925
  Injection-site reactions: Week 4 | 9.6 (0.7)
  Injection-site reactions: Week 8: number analyzed (Participants) | 907
  Injection-site reactions: Week 8 | 9.6 (0.8)
  Injection-site reactions: Week 12: number analyzed (Participants) | 862
  Injection-site reactions: Week 12 | 9.6 (0.7)
  Injection-site reactions: Week 24: number analyzed (Participants) | 679
  Injection-site reactions: Week 24 | 9.5 (0.9)
  Injection-site reactions: Week 48: number analyzed (Participants) | 549
  Injection-site reactions: Week 48 | 9.5 (0.8)
  Injection-site reactions: Week 72: number analyzed (Participants) | 431
  Injection-site reactions: Week 72 | 9.5 (0.8)
  Injection-site reactions: Week 96: number analyzed (Participants) | 353
  Injection-site reactions: Week 96 | 9.5 (0.8)
  Ease of use: Week 4: number analyzed (Participants) | 927
  Ease of use: Week 4 | 8.7 (1.5)
  Ease of use: Week 8: number analyzed (Participants) | 914
  Ease of use: Week 8 | 8.7 (1.6)
  Ease of use: Week 12: number analyzed (Participants) | 866
  Ease of use: Week 12 | 8.8 (1.6)
  Ease of use: Week 24: number analyzed (Participants) | 676
  Ease of use: Week 24 | 8.8 (1.6)
  Ease of use: Week 48: number analyzed (Participants) | 559
  Ease of use: Week 48 | 8.9 (1.4)
  Ease of use: Week 72: number analyzed (Participants) | 432
  Ease of use: Week 72 | 9.0 (1.5)
  Ease of use: Week 96: number analyzed (Participants) | 353
  Ease of use: Week 96 | 9.0 (1.4)

ADVERSE EVENTS:
Time Frame: All AEs were collected from first injection of IMP up to 2 weeks after last dose of study drug (Week 120).
Description: Reported AEs and deaths were TEAEs that developed or worsened or became serious and deaths that occurred during the TEAE period (time from the first injection of study drug up to the day of the last injection of study drug + 14 days). Analysis was performed on safety population.
Arm/Group | Alirocumab
All-Cause Mortality (participants affected / at risk) | 2/994
Serious Adverse Events (participants affected / at risk) | 161/994
Other Adverse Events (participants affected / at risk) | 221/994
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alirocumab (N=994)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Acute Coronary Syndrome (Cardiac disorders) | 5 (5)
Acute Myocardial Infarction (Cardiac disorders) | 5 (5)
Angina Pectoris (Cardiac disorders) | 15 (15)
Angina Unstable (Cardiac disorders) | 12 (14)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 5 (5)
Atrial Flutter (Cardiac disorders) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular Block Second Degree (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 3 (3)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 6 (6)
Coronary Artery Stenosis (Cardiac disorders) | 6 (7)
Coronary Ostial Stenosis (Cardiac disorders) | 1 (1)
Mitral Valve Stenosis (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Myocardial Ischaemia (Cardiac disorders) | 5 (5)
Subendocardial Ischaemia (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Accessory Navicular Syndrome (Congenital, familial and genetic disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Perianal Erythema (Gastrointestinal disorders) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Vascular Stent Stenosis (General disorders) | 4 (4)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Chronic Hepatitis (Hepatobiliary disorders) | 1 (1)
Hepatocellular Injury (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Campylobacter Colitis (Infections and infestations) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3)
Escherichia Sepsis (Infections and infestations) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 2 (2)
Liver Abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 2 (3)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 2 (2)
Scapula Fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal Column Injury (Injury, poisoning and procedural complications) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 3 (3)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 (2)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 (1)
Transaminases Increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 (3)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign Neoplasm Of Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Cancer Stage 0, With Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 3 (3)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Facial Paralysis (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 3 (3)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Device Dislocation (Product Issues) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Schizophrenia (Psychiatric disorders) | 1 (1)
Bladder Trabeculation (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pregnancy Of Partner (Social circumstances) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Aortic Dissection (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 2 (2)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1)
Peripheral Artery Stenosis (Vascular disorders) | 2 (2)
Peripheral Artery Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alirocumab (N=994)
Influenza (Infections and infestations) | 53 (61)
Nasopharyngitis (Infections and infestations) | 78 (86)
Myalgia (Musculoskeletal and connective tissue disorders) | 71 (93)
Headache (Nervous system disorders) | 61 (94)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02476006/Prot_001.pdf
  • Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT02476006/SAP_000.pdf